CLINICAL TRIAL: NCT05304884
Title: Clinical and Functional Outcomes of a Single Dose Ozone, Three Doses of Ozone and Corticosteroid Injection in Patients With Shoulder Impingement Syndrome
Brief Title: Ozone Injection for Shoulder Impengement Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Mehmet Cenk Turgut, MD, Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/11/177
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Research on the Effectiveness of a Corticosteroid, Single Dose and Three Doses of Ozone Injection in Shoulder Impingement Syndrome
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Group 1 received a single dose (n:36), group 2 (n:36) received three doses of ozone injection (n :36). Group 3 (n:36) was treated with a corticosteroid injection.
Who Masked: Outcomes Assessor
Masking Description: Interventions were perfored by a physician and study outcomes were assessed by another physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single dose ozone (Active Comparator): Group 1 received a single dose ozone injection (n:36)
  Interventions: Combination Product: combined oxygen-ozone and corticosteroid
- three doses of ozone (Active Comparator): Group 2 (n:36) received three doses of ozone injection (n :36).
  Interventions: Combination Product: combined oxygen-ozone and corticosteroid
- corticosteroid (Active Comparator): Group 3 (n:36) was treated with a corticosteroid injection
  Interventions: Combination Product: combined oxygen-ozone and corticosteroid

INTERVENTIONS:
Combination Product: combined oxygen-ozone and corticosteroid — Subacromial injection using Ultrasound

SUMMARY:
Ozone injection has lately been utilized as a safe alternative to corticosteroids in the management of musculoskeletal diseases with fewer side effects. This study aimed to compare the effectiveness of a corticosteroid, single dose and three doses of ozone injection in shoulder impingement syndrome (SIS).

DETAILED DESCRIPTION:
A hundred and eight SIS patients were divided into three groups and underwent subacromial injections in this prospective study. Group 1 received a single dose (n:36), group 2 (n:36) received three doses of ozone injection (n :36). Group 3 (n:36) was treated with a corticosteroid injection. Patients were evaluated using the visual analog scale (VAS) and Constant Murley Score (CMS), pre-injection and at 4 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria: patients older than 18 years with shoulder pain lasting for more than three months, pain severity more than 5/10 on Visual Analog Scale (VAS), and diagnosed with SIS according to clinical examination and magnetic resonance imaging (MRI), were enrolled in this randomized clinical study.

-

Exclusion Criteria: The exclusion criteria were as follows: existing pathological abnormalities such as full-thickness rotator cuff tears on MRI, any cause of shoulder pain other than SIS such as inflammatory joint diseases, shoulder osteoarthritis and adhesive capsulitis, restriction of shoulder range of motion, coagulation disorders or use of anticoagulants, previous history of shoulder trauma, surgery or fracture, history of any subacromial injection or physical therapy for the last year, contraindications for ozone injection such as known Glucose 6 phosphate dehydrogenase deficiency, pregnancy, uncontrolled hyperthyroidism, and leukemia.

-

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
The visual analog scale (VAS) | 3 months

SECONDARY OUTCOMES:
Constant Murley Score (CMS) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- KTU Medical Faculty, Merkez, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided